CLINICAL TRIAL: NCT04217083
Title: Volatile Organic Compounds (VOCs) Could Discriminate Patients With Colorectal Cancer From Healthy Controls.
Brief Title: Volatile Organic Compounds (VOCs) Profile in Colorectal Cancer Patients and Healthy Controls.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Sponsor
Other Study IDs: 141/2019
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer; Colon Polyp
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal cancer patients: Patients with histologically proven Colorectal cancer detected during the colonoscopy
  Interventions: Diagnostic Test: Breath sampling
- healthy controls: Patients with no sign of any colorectal disease who are submitted to colonoscopy
  Interventions: Diagnostic Test: Breath sampling

INTERVENTIONS:
Diagnostic Test: Breath sampling — The alveolar fraction of Colorectal cancer patients and Healthy controls will be sampled using a breath sampler able to fix the volatile organic compound on absorbable tubes

SUMMARY:
Volatile organic compounds (VOCs) are low molecular weight (<1 kDa) compounds which represent the final products of cell metabolism. Their composition can be affected by several factors including diet, hormones, environment and the presence of diseases, in particular, cancer.

Colorectal cancer (CRC) is one of the commonest tumours and is an important cause of cancer-related mortality.

The expression of VOCs in breath that are linked to a patient's disease state could offers a powerful, non-invasive approach to identifying CRC patients.

DETAILED DESCRIPTION:
Volatile organic compounds (VOCs) are low molecular weight (<1 kDa) compounds which represent the final products of cell metabolism. Their composition can be affected by several factors including diet, hormones, environment and the presence of diseases, in particular, cancer.

Endogenous breath VOCs can originate anywhere in the body, reversed in the venous blood stream and than to the lung alveoli where some of them are exhaled .

Alteration in VOC production in patients with cancer has been postulated to relate to (per)oxygenation of cell membrane-based polyunsaturated fatty acids resulting from genetic and/or protein mutations within tumour cells and the increased relative prevalence of reactive oxygen species within cancer cells. VOCs consist largely of benzene, alkanes and aldehydes (or their derivatives), and several studies have demonstrated that various cancers, including lung and breast cancer,melanoma, mesothelioma and hepatocellular carcinoma, are associated with specific VOC profiles that differ from normal.

Volatile organic compounds are present in various excreted biological materials (urine, blood, faeces an breath) and their analysis offers a possibility for cancer screening.

Colorectal cancer (CRC) is one of the commonest tumours and is an important cause of cancer-related mortality. It is the second leading cause of cancer-related death in Europe and the third in the USA.

Colonoscopy is the gold standard for the diagnosis of CRC, although its cost prevents its use for mass screening. Furthermore colonoscopy is not well accepted by patients since it is an invasive exam. Faecal immunochemical blood testing (FIT) is the most widely used noninvasive screening tool, showing fairly good specificity but a high variation in sensitivity (61-91%) and adherence to screening programmes rarely reaches 50-70% of the target population.

The expression of VOCs in breath that are linked to a patient's disease state could offers a powerful, non-invasive approach to identifying CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 95
* Histologically proven colorectal cancer
* Patient with single or multiple polyps of the colon
* Healthy subjects with negative colonoscopy
* Patients already sampled and operated for colorectal cancer with no sign of recurrence
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Inflammatory bowel disease
* Synchronous cancers
* Liver and/or lung metastasis
* Bowel prep
* Recurrent CRC
* Any psychiatric disease
* Emergency operations

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients which will be consulted at the Tertiary center of colorectal surgery (Policlinico of Bari)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-25 (Estimated); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
Test Sensitivity and specificity for colorectal cancer | 30 days
  A specificity of 80% and a sensitivity of 90% will be considered reliable

SECONDARY OUTCOMES:
Test Sensitivity and specificity for colorectal polyps | 30 days
  A specificity of 80% and a sensitivity of 90% will be considered reliable

CONTACTS AND LOCATIONS:
Overall Officials: Donato Altomare, Prof, Principal Investigator — Societa Italiana di Chirurgia ColoRettale
Locations (1):
- Dept of Emergency and Organ transplantation - University of Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fuchs P, Loeseken C, Schubert JK, Miekisch W. Breath gas aldehydes as biomarkers of lung cancer. Int J Cancer. 2010 Jun 1;126(11):2663-70. doi: 10.1002/ijc.24970. PMID 19839051
- [Result] Bond A, Greenwood R, Lewis S, Corfe B, Sarkar S, O'Toole P, Rooney P, Burkitt M, Hold G, Probert C. Volatile organic compounds emitted from faeces as a biomarker for colorectal cancer. Aliment Pharmacol Ther. 2019 Apr;49(8):1005-1012. doi: 10.1111/apt.15140. Epub 2019 Mar 3. PMID 30828825
- [Result] Arasaradnam RP, McFarlane MJ, Ryan-Fisher C, Westenbrink E, Hodges P, Thomas MG, Chambers S, O'Connell N, Bailey C, Harmston C, Nwokolo CU, Bardhan KD, Covington JA. Detection of colorectal cancer (CRC) by urinary volatile organic compound analysis. PLoS One. 2014 Sep 30;9(9):e108750. doi: 10.1371/journal.pone.0108750. eCollection 2014. PMID 25268885
- [Result] Altomare DF, Di Lena M, Porcelli F, Trizio L, Travaglio E, Tutino M, Dragonieri S, Memeo V, de Gennaro G. Exhaled volatile organic compounds identify patients with colorectal cancer. Br J Surg. 2013 Jan;100(1):144-50. doi: 10.1002/bjs.8942. PMID 23212621